CLINICAL TRIAL: NCT04322734
Title: Transgenerational Metabolic-Immune Biomarkers of Neurological and Neurodevelopmental Disorders
Status: Recruiting | Type: Observational
Sponsor: Southwest Autism Research & Resource Center (Other)
Collaborators: State University of New York - Downstate Medical Center (Other)
Responsible Party: Principal Investigator, Richard Frye, Principal Investigator and Sponsor, Southwest Autism Research & Resource Center
Other Study IDs: Mito Tissue
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Autism Spectrum Disorder; Mitochondrial Pathology; Epilepsy; Brain Tumor; Psychiatric Disorder; Mitochondrial Diseases
MeSH Terms: conditions — Autism Spectrum Disorder; Epilepsy; Brain Neoplasms; Mental Disorders; Mitochondrial Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will examine multiple aspects of metabolic disorders in tissue, blood and cerebrospinal fluid in patient with brain based disorders, typically developing siblings and biological parents. Genetic and epigenetic markers will be examined in blood and/or saliva. Baby teeth, hair, medical history and resident location will be analyzed to assess environmental exposures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- ASD (General): 150 children with ASD and unknown MD status
- ASD (With MD): 50 children with ASD and confirmed MD
- ASD (No MD): 50 children with ASD and ruled out MD
- Epilepsy: 50 children with epilepsy (primary) and no ASD
- Brain Tumor: 50 children with brain tumor (primary) and no ASD
- Psychiatric Disorder: 50 children with psychiatric disorder (primary) and no ASD, using lithium treatments
- MD (No ASD): 50 children with MD (primary) and no ASD
- TD (With ASD Sibling): 50 TD children with a sibling with ASD/neurodevelopmental delay
- TD (No ASD Sibling): 50 TD children with no siblings with ASD/neurodevelopmental delay

SUMMARY:
The study involves up to 5 visits for a fasting blood draw, behavioral assessments, and/or questionnaires. Other samples may be collected when appropriate.

This study is currently recruiting.

There is no cost for visits or study-related exams.

DETAILED DESCRIPTION:
Mitochondria are essential for a wide range of functions in almost every cell in our body. Best known for their role in adenosine triphosphate (ATP) production, mitochondria are also closely involved in a wide variety of cell functions such as calcium buffering, redox regulation, apoptosis and inflammation, and regulate metabolism through several mechanisms, including epigenetic changes. ATP produced is essential for many cellular systems. Thus, abnormal mitochondrial function can adversely affect cellular systems by several mechanisms.

Given the important role of the mitochondria in cellular function, individuals with classic mitochondrial disease demonstrate devastating symptoms, particularly in tissues that have high-energy demands such as the brain, muscles, gastrointestinal (GI) tract and immune system. Mitochondrial dysfunction contributes to the pathophysiology of more common diseases, including psychiatric diseases, neurodegenerative disorders, neurological disorders including migraine and seizures, persistent systemic inflammation, cardiac disease, cancer and diabetes. Mitochondrial dysfunction also effects a significant portion of individuals with autism spectrum disorder (ASD) as well as genetic syndromes associated with ASD.

One of our goals is to develop a method using the Seahorse Analyzer to measure individual variations in mitochondrial function which can identify children with medical disorders and mitochondrial dysfunction without an invasive muscle biopsy. In order to establish comprehensive profiles of mitochondrial function for individuals with known neurological and neurodevelopmental disorders, we will compare blood, urine, and stool from these individuals to those of healthy, typically developing (TD) children. The relationship between mitochondrial function, development, and behavior will be assessed by performing standard developmental testing. In addition, in patients who have a procedure that produces leftover tissue, we will examine the mitochondrial function in that tissue and correlate it with findings from blood.

ELIGIBILITY:
Inclusion Criteria (ASD):

1. ASD, as defined by either a gold standard measure for ASD diagnosis, the Autism Diagnostic Observation Schedule (ADOS); the Autism Diagnostic Interview-Revised (ADI-R); and/or a comprehensive assessment that is consistent with ASD, in the opinion of the principal investigator. For those the PI believes a prospective diagnosis of ASD is warranted, a formal diagnostic assessment will be scheduled at screening.
2. 0 years through 17 years 11 months of age

Inclusion Criteria (TD, MD, Epilepsy, Brain Tumor, Psychiatric)

1. 0 years to 17 years 11 months of age

Exclusion Criteria (All):

1. History of a significant adverse reaction to a prior blood draw
2. In females of reproductive age, pregnancy or plans to become pregnant
3. Any other historical event/information that may, in the opinion of the PI, be a reason to exclude the child from participation.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 400 children aged 0 years to 17 years 11 months with a neurological, psychiatric or neurodevelopmental disorder.
  250 children in this sample will have a known diagnosis of ASD: 50 children with a diagnosed MD (ASD/MD), 50 children with ruled out MD (ASD/NoMD), 150 children with ASD and unknown MD status.
  Comparison groups: 50 children with epilepsy (without ASD), 50 with psychiatric disorders, 50 with brain tumors (without ASD) 50 with a diagnosed MD (without ASD)
  Control group: 100 TD children (50 siblings of children with ASD and 50 without any siblings with ASD or developmental delay).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Mitochondrial Reserve Capacity measured using the Seahorse XR Flux Analyzer | Up to one year
  Children with ASD will be differentiated from all other cohorts and have a specific pattern of mitochondrial dysfunction that will be different from and comparable to other groups of children in the study (e.g. mitochondrial disease without autism, typically developing, autism with mitochondrial disease, and developmental delay). It is hypothesized that these children will have a more pronounced delay in their development and will have a higher probability for poor developmental and behavioral outcomes. This will be evaluated using a Seahorse XR flux analyzer to generate a maximal reserve capacity value.

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Frye, MD, PhD, Study Director — Autism Discovery & Treatment Foundation
Locations (2):
- United States (2):
  - Southwestern Research and Resource Center, Phoenix, Arizona
  - State University of New York, Downstate, Brooklyn, New York

IPD SHARING:
Plan to Share IPD: Yes
The PI may collaborate with other researchers to perform analyses on individual samples that have been stored for future research. In this case, the coded data with characteristics about the participant will be shared as appropriate (e.g., diagnostic status).
Time Frame: After completion of initial study
Access Criteria: Researchers must have an established protocol with relevant interest to the samples and data stored.